CLINICAL TRIAL: NCT04633343
Title: Effects of Different Tidal Volume Ventilation Strategies on Fontan Flow and Hemodynamics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Manchula Navaratnam, Clinical Associate Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 58526
Record Dates: First submitted 2020-11-11; First posted 2020-11-18 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2023-05

CONDITIONS: Fontan Physiology

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Small Volume Breath Group (5mlKg) (Experimental): Small volume breath and fast breathing rate for 5 minutes when the patient is in the Operating room and on mechanical ventilation
  Interventions: Other: Small volume breath and fast breathing rate for 5 minutes
- Large Volume Breath Group (10mL/kg) (Experimental): Large volume breath and slow breathing rate for 5 minutes when the patient is in the Operating room and on mechanical ventilation.
  Interventions: Other: Large volume breath and slow breathing rate for 5 minutes

INTERVENTIONS:
Other: Small volume breath and fast breathing rate for 5 minutes — Small volume breath and fast breathing rate delivered via mechanical ventilator.
  Arms: Small Volume Breath Group (5mlKg)
Other: Large volume breath and slow breathing rate for 5 minutes — Large volume breath and slow breathing rate delivered via mechanical ventilator.
  Arms: Large Volume Breath Group (10mL/kg)

SUMMARY:
In patients with Fontan circulation blood is not pumped to the lungs from a ventricle. Instead the superior vena cava and inferior vena cava is connected to the pulmonary artery and blood flow to the lungs occurs passively along this Fontan pathway. This passive blood flow to the lungs occurs best when the patient is breathing on their own (spontaneous ventilation). However for certain surgeries and procedures patients need to have an endotracheal tube inserted and need to be muscle relaxed and receive positive pressure ventilation. Prior studies have shown that positive pressure ventilation can reduce blood flow to the lungs and consequently blood returning to the heart resulting in less blood pumped out to the rest of the body (cardiac output). The purpose of this study is to investigate if changing the volume of the positive pressure ventilation (tidal volume) affects blood flow to the lungs and cardiac output in patients with Fontan circulation.

DETAILED DESCRIPTION:
If it can be shown that changing the tidal volume does affect the blood flow to the lungs and cardiac output in patients with Fontan circulation the information can be used to learn from this study to optimize the tidal volume ventilation, and therefore pulmonary blood flow and cardiac output when Fontan patients come for general anesthesia. This is important because the population of patients with Fontan circulation is increasing and an increasing number will present for cardiac and non cardiac surgery when positive pressure ventilation will be required. They may also spend time on the cardiac intensive care unit on a ventilator and improving our knowledge on how best to ventilate them may help improve their overall hospital outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Age 2- 50 years of age
2. Patients with Fontan circulation undergoing cardio-thoracic surgery or undergoing cardio-thoracic surgery for completion of Fontan circulation.

Exclusion Criteria:

1. Patients presenting for cardio-thoracic surgery without Fontan circulation or those not coming for completion of Fontan circulation.

Ages: 2 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2021-02-22 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Transpulmonary gradient | 5 minutes of change in Tidal Volume (high vs low)
  Effect of tidal volume changes (high vs low) on Transpulmonary gradient as measured as the difference between mean pulmonary artery pressure measured from right internal jugular (Fontan pressure line) and left atrial pressure measured by direct intracardiac pressure line. Both lines are placed for the scheduled clinical procedure and not solely for the purposes of the research study.

SECONDARY OUTCOMES:
Blood flow in inferior vena cava (IVC) | 5 minutes of change in Tidal Volume (high vs low)
  Effect of tidal volume changes (high vs low) on blood flow in inferior vena cava (IVC) as measured by Transesophageal Echocardiography TEE)..
Systemic outflow tract stroke distance (velocity time integral) | 5 minutes of change in Tidal Volume (high vs low)
  Effect of tidal volume changes (high vs low) on systemic outflow tract stroke distance (velocity time integral) as measured by Transesophageal Echocardiography. (TEE).

CONTACTS AND LOCATIONS:
Overall Officials: Manchula Navaratnam, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Navaratnam M, Schmidt AR, Kaplinski M, De Souza E, Beattie MJ, Rowe EV, Punn R, Ramamoorthy C. Hemodynamic Effects of Altering Tidal Volume During Positive Pressure Ventilation in the Fontan Circulation: A Randomized Crossover Trial. Paediatr Anaesth. 2025 Aug;35(8):607-618. doi: 10.1111/pan.15096. Epub 2025 Mar 19. PMID 40105302